CLINICAL TRIAL: NCT02446015
Title: Clinical Evaluation Following Use of SYSTANE® ULTRA in the Management of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXC120-P001
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systane Ultra QID (Experimental): SYSTANE® ULTRA lubricant eye drops,1 drop in each eye, 4 times per day (QID) for 28 days
  Interventions: Drug: SYSTANE® ULTRA Lubricant Eye Drops
- Systane Ultra PRN (Active Comparator): SYSTANE® ULTRA lubricant eye drops, 1 drop in each eye, as needed (PRN) for 28 days
  Interventions: Drug: SYSTANE® ULTRA Lubricant Eye Drops

INTERVENTIONS:
Drug: SYSTANE® ULTRA Lubricant Eye Drops
  Other Names: SYSTANE® ULTRA

SUMMARY:
The purpose of this study is to evaluate the clinical benefits of SYSTANE® ULTRA Lubricant Eye Drops using total ocular surface staining scores in subjects with dry eye administering it either as a scheduled regimen or as-needed after 28 days of treatment.

DETAILED DESCRIPTION:
This study consists of a 14-day Run-in Phase (between the Screening Visit and Baseline/Visit 1) and a Treatment Phase. During the Run-in Phase, subjects will discontinue current artificial tears and will be dispensed SYSTANE® ULTRA to be administered 1 drop in each eye as needed (PRN). Subjects who meet the re-evaluation criteria after the Run-in Phase will be randomized in a 1:2 manner to receive treatment with SYSTANE® ULTRA 4 times per day (QID) or PRN, respectively, for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend all study visits.
* Use of BAK-free artificial tear drops on an as needed basis, at least once a week, for at least 3 months prior to Screening Visit (maximum use of 4 drops a day).
* At least one '8 hour waking period' per week during the run-in phase without using the provided artificial tear.
* Use provided artificial tear at least once a week during run-in phase.
* Willing to take study treatment as directed for the entire study and able to complete the study diaries as required.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Use of artificial tears, as specified in the protocol.
* Use of topical ocular medications, as specified in the protocol.
* Women of childbearing potential who are pregnant, breast feeding, plan to become pregnant during the study, or not using adequate birth control methods to prevent pregnancy throughout the study.
* Any hypersensitivity to the use of the study product formulations or an allergy to any ingredient(s) contained within product formulations.
* Ocular abnormalities, infection, or active inflammation (not associated with dry eye) as specified in the protocol.
* Ocular or intraocular surgery or serious ocular trauma in either eye within the past 6 months prior to Screening Visit.
* Any medical condition (systemic or ophthalmic) that may preclude the safe administration of test article or safe participation in the study.
* Contact lens use within 2 weeks prior to Screening Visit, and unwilling to avoid contact lens use during the course of the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Study Director — Alcon Research

REFERENCES:
- [Derived] Asbell P, Vingrys AJ, Tan J, Ogundele A, Downie LE, Jerkins G, Shettle L. Clinical Outcomes of Fixed Versus As-Needed Use of Artificial Tears in Dry Eye Disease: A 6-Week, Observer-Masked Phase 4 Clinical Trial. Invest Ophthalmol Vis Sci. 2018 May 1;59(6):2275-2280. doi: 10.1167/iovs.17-23733. PMID 29715369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study centers located in the US and 2 study centers located in Australia.
Pre-assignment Details: Of the 159 enrolled, 58 subjects were exited as screen failures prior to randomization. An additional 4 subjects were randomized in error and did not receive investigational product (IP). This reporting group includes all treated subjects (97).
Period: Overall Study
Arm/Group | Systane Ultra QID | Systane Ultra PRN
Started | 34 | 63
Completed | 33 | 62
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received at least 1 dose of the randomized investigational product (Intent-to-Treat Analysis Set).
Groups:
- Systane Ultra QID: SYSTANE® ULTRA lubricant eye drops,1 drop in each eye QID for 28 days
- Systane Ultra PRN: SYSTANE® ULTRA lubricant eye drops, 1 drop in each eye PRN for 28 days
- Total: Total of all reporting groups
Arm/Group | Systane Ultra QID | Systane Ultra PRN | Total
Number analyzed (Participants) | 34 | 63 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (16.6) | 52.2 (18.1) | 50.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 51 | 77
  Male | 8 | 12 | 20
Total Ocular Surface Staining (TOSS) Score [Mean (Standard Deviation); unit: units on a scale] — The TOSS score is a cumulative cornea and conjunctival staining score. After instilling ophthalmic dye in the eye, the investigator graded three areas of the ocular surface for dryness on a scale from 0 to 5, where 0 is "Absent" and 5 is "Severe." The three scores were summed for a resultant overall 0-15 score.
  units on a scale | 5.1 (1.28) | 5.0 (1.07) | 5.0 (1.14)
Impact of Dry Eye on Everyday Life Symptom-Bother (IDEEL SB) Score [Mean (Standard Deviation); unit: units on a scale] — The IDEEL SB module is a 20 question patient reported outcome questionnaire that assesses the subject's symptoms of dry eye. An overall resultant calculated score ranges from 0 to 100, with higher scores indicating greater symptom bother.
  units on a scale | 43.20 (11.049) | 46.75 (9.854) | 45.50 (10.372)
IDEEL Treatment Satisfaction Scores [Mean (Standard Deviation); unit: units on a scale] — The IDEEL is 10-question patient-reported outcome questionnaire that assesses the subject's general satisfaction with treatment use (Treatment Effectiveness and Treatment Inconvenience). A resultant overall 0-100 treatment satisfaction score was calculated separately for Treatment Effectiveness and Treatment Inconvenience, with higher scores indicating greater satisfaction and less treatment-related bother.
  units on a scale
    Effectiveness | 57.17 (20.708) | 57.54 (20.428) | 57.41 (20.419)
    Inconvenience | 84.38 (15.329) | 84.03 (14.189) | 84.15 (14.520)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Ocular Surface Staining (TOSS) Score at Day 28
Description: The TOSS score is a cumulative cornea and conjunctival staining score. After instilling ophthalmic dye in the eye, the investigator graded three areas of the ocular surface for dryness on a scale from 0 to 5, where 0 is "Absent" and 5 is "Severe." The three scores were summed for a resultant overall 0-15 score. The change from baseline was calculated as the TOSS score at Day 28 minus the TOSS score at baseline. A more negative change value indicates greater efficacy. One eye from each subject was chosen as the study eye and only the study eye was used for eye-level efficacy analyses.
Time Frame: Baseline (Day 0), Day 28
Population: Intent-to-Treat Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Ultra QID | Systane Ultra PRN
Number analyzed (Participants) | 33 | 62
units on a scale | -1.19 (0.26) | -0.94 (0.24)

2. Secondary Outcome: Change From Baseline in Impact of Dry Eye on Everyday Life Symptom-Bother (IDEEL SB) Score at Day 28
Description: The IDEEL SB module is a 20 question patient reported outcome questionnaire that assesses the subject's symptoms of dry eye. An overall resultant calculated score ranges from 0 to 100, with higher scores indicating greater symptom bother. One eye from each subject was chosen as the study eye and only the study eye was used for eye-level efficacy analyses.
Time Frame: Baseline (Day 0), Day 28
Population: Intent-to-Treat Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Ultra QID | Systane Ultra PRN
Number analyzed (Participants) | 33 | 62
units on a scale | -7.00 (2.01) | -2.94 (1.85)

3. Secondary Outcome: Change From Baseline in IDEEL Treatment Satisfaction Scores (Treatment Effectiveness and Treatment-related Inconvenience) at Day 28
Description: The IDEEL is 10-question patient-reported outcome questionnaire that assesses the subject's general satisfaction with treatment use (Treatment Effectiveness and Treatment Inconvenience). A resultant overall 0-100 treatment satisfaction score was calculated separately for Treatment Effectiveness and Treatment Inconvenience, with higher scores indicating greater satisfaction and less treatment-related bother. One eye from each subject was chosen as the study eye and only the study eye was used for eye-level efficacy analyses.
Time Frame: Baseline (Day 0), Day 28
Population: Intent-to-Treat Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Ultra QID | Systane Ultra PRN
Number analyzed (Participants) | 33 | 62
units on a scale
  Effectiveness | 2.43 (3.53) | 0.16 (3.21)
  Inconvenience | -11.56 (2.94) | -2.77 (2.67)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 6 weeks). AEs are reported as pre-treatment and treatment-emergent
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from participants and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- Systane Ultra QID: All subjects treated with SYSTANE® ULTRA lubricant eye drops QID
- Systane Ultra PRN: All subjects treated with SYSTANE® ULTRA lubricant eye drops PRN
Arm/Group | Pretreatment | Systane Ultra QID | Systane Ultra PRN
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/34 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/34 | 0/63
Other Adverse Events (participants affected / at risk) | 0/159 | 0/34 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.